CLINICAL TRIAL: NCT05794477
Title: An Open Label, Multicenter, Phase Ib/II Study of SHR-1802 in Combination With Adebrelimab in Patients With Advanced Solid Tumors
Brief Title: A Study of SHR-1802 in Combination With Adebrelimab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1802-II-202
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Carboplatin; Cisplatin; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Dose-exploration：Six patients will be enrolled for tolerability observation. If ≥2 subjects in the previous dose level experienced DLTS, an additional 6 subjects in the other dose level were enrolled.
  Efficacy-expansion: After determination of the recommended dose for Phase II (RP2D), selected cohorts with different tumor types will be expanded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- phase Ib：SHR-1802+Adebrelimab (Experimental)
  Interventions: Biological: Adebrelimab; Biological: SHR-1802
- phase II cohort 1: SHR-1802+Adebrelimab (Experimental)
  Interventions: Biological: Adebrelimab; Biological: SHR-1802
- phase II cohort 2: SHR-1802+Adebrelimab + Platinum Doublet Chemotherapy (PDCT) (Experimental)
  Interventions: Biological: Adebrelimab; Biological: SHR-1802; Drug: Carboplatin/Cisplatin; Drug: Paclitaxel/Nab-Paclitaxel/Pemetrexed
- phase II cohort 3: SHR-1802+Adebrelimab + PDCT (Experimental)
  Interventions: Biological: Adebrelimab; Biological: SHR-1802; Drug: Carboplatin/Cisplatin; Drug: Paclitaxel/Nab-Paclitaxel/Pemetrexed
- phase II cohort 4: SHR-1802+Adebrelimab (Experimental)
  Interventions: Biological: Adebrelimab; Biological: SHR-1802

INTERVENTIONS:
Biological: Adebrelimab — Specified dose on specified days
Biological: SHR-1802 — Specified dose on specified days
Drug: Carboplatin/Cisplatin — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
  Arms: phase II cohort 2: SHR-1802+Adebrelimab + Platinum Doublet Chemotherapy (PDCT); phase II cohort 3: SHR-1802+Adebrelimab + PDCT
Drug: Paclitaxel/Nab-Paclitaxel/Pemetrexed — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
  Arms: phase II cohort 2: SHR-1802+Adebrelimab + Platinum Doublet Chemotherapy (PDCT); phase II cohort 3: SHR-1802+Adebrelimab + PDCT

SUMMARY:
The aim of this study is to observe and evaluate the tolerability, safety, pharmacokinetics and immunogenicity of SHR-1802 combined with adebrelimab in patients with advanced solid tumors, determine the RP2D of SHR-1802 combined with adebrelimab ± chemotherapy, and evaluate the efficacy of SHR-1802 combined with adebrelimab ± chemotherapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Has a life expectancy≥ 12 weeks；
4. At least one measurable lesion according to RECIST v1.1；
5. Pathologically confirmed advanced solid tumor；
6. Adequate bone marrow reserve and organ function.

Exclusion Criteria:

1. Have received anti-PD-1 or PD-L1 antibody therapy;
2. Subjects with other malignant tumors in the past 3 years;
3. Have uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites;
4. Previous or current interstitial pneumonia/interstitial lung disease ;
5. History of autoimmune disease with the possibility of recurrence or active autoimmune disease;
6. Severe infection within 1 month before the first study drug administration;
7. The presence of other serious physical or mental disorders or abnormalities in laboratory tests that may increase the risk of study participation or interfere with study results, as well as patients deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 3 weeks
Recommended phase II dose (RP2D) | up to 2 months
ORR | up to 2 years
  Objective Response Rate, determined according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
DOR | up to 2 years
  Duration of Response, determined according to RECIST v1.1 criteria
DCR | up to 2 years
  Disease Control Rate, determined according to RECIST v1.1 criteria
PFS assessed by investigator | up to 2 years
  Progression Free Survival, determined according to RECIST v1.1 criteria
TTR | up to 2 years
  Time to Response，determined according to RECIST v1.1 criteria
OS (overall survival) | up to 2 years
  From date of treatment start to any cause death or last follow-up
12-month OS rate | from the date of the first dose up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided